CLINICAL TRIAL: NCT00022529
Title: Phase I Study of Intravenous BMS-214662 FTI (NSC# 710086) and Herceptin (NSC# 688097) Weekly in Patients With Advanced Malignancies
Brief Title: BMS-214662 Plus Trastuzumab in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02396; FCCC-01013; CDR0000068828 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-08-10; First posted 2003-06-17 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — 7-cyano-2,3,4,5-tetrahydro-1-(1H-imidazol-4-ylmethyl)-3-(phenylmethyl)-4-(2-thienylsulfonyl)-1H-1,4-benzodiazepine; Trastuzumab

ARMS (1):
- Treatment (BMS-214662, trastuzumab) (Experimental): Patients receive BMS-214662 IV over 1 hour on days 2, 8, 15, and 22 and trastuzumab (Herceptin) IV over 30-90 minutes on days 1, 8, 15, and 22. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: BMS-214662; Biological: trastuzumab; Other: pharmacological study

INTERVENTIONS:
Drug: BMS-214662 — Given IV
  Other Names: farnesyltransferase inhibitor BMS-214662; FTI BMS 214662
Biological: trastuzumab — Given IV
  Other Names: anti-c-erB-2; Herceptin; MOAB HER2
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Phase I trial to study the effectiveness of BMS-214662 plus trastuzumab in treating patients who have advanced solid tumors. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Combining monoclonal antibody therapy with chemotherapy may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose and recommended phase II dose of BMS-214662 when combined with trastuzumab (Herceptin) in patients with advanced solid tumors.

II. Determine the dose-limiting toxic effects of this regimen in these patients.

SECONDARY OBJECTIVES:

I. Determine the pharmacokinetics of this regimen in these patients. Ii. Determine, in a preliminary manner, the antitumor activity of this regimen in these patients.

OUTLINE: This is a dose-escalation study of BMS-214662.

Patients receive BMS-214662 IV over 1 hour on days 2, 8, 15, and 22 and trastuzumab (Herceptin) IV over 30-90 minutes on days 1, 8, 15, and 22. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of BMS-214662 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are accrued to receive treatment with BMS-214662 and trastuzumab at the recommended phase II dose.

PROJECTED ACCRUAL: A total of 3-28 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed solid tumor that is unresponsive to currently available therapies or for which no known effective therapy exists
* Overexpressing HER-2-neu (2+ or 3+) by immunohistochemistry or fluorescent in situ hybridization
* Clinically or radiologically evaluable disease
* No carcinomatous meningitis or untreated/uncontrolled metastatic brain parenchymal disease

  * At least 8 weeks since prior therapy for prior brain parenchymal disease and asymptomatic off corticosteroids
* Performance status - ECOG 0-2
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.8 mg/dL
* ALT and AST no greater than 1.5 times upper limit of normal (ULN)
* Creatinine no greater than 1.5 times ULN
* No uncontrolled or significant cardiovascular disease
* No myocardial infarction within the past 6 months
* No prior clinically significant atrial or ventricular arrhythmias
* No prior second or third degree heart block
* No ischemic heart disease requiring medication
* No congestive heart failure
* Corrected QT interval no greater than 450 milliseconds by electrocardiogram
* Ejection fraction at least lower limit of normal by MUGA scan
* No uncontrolled or significant pulmonary disease
* No active unresolved infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study
* At least 4 weeks since prior immunotherapy, including trastuzumab (Herceptin), and recovered
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No anthracyclines for at least 22 weeks after completion of study therapy
* No other concurrent chemotherapy
* Concurrent hormone replacement therapy allowed
* No other concurrent hormonal therapy
* At least 4 weeks since prior radiotherapy and recovered
* No prior radiotherapy to more than 25% of the bone marrow-containing skeleton
* No concurrent radiotherapy
* At least 4 weeks since prior investigational agents and recovered
* At least 7 days since prior known substrates of cytochrome P450-3A4 (CYP3A4)
* At least 7 days since prior parenteral antibiotics
* No concurrent substrates of CYP3A4
* No concurrent parenteral antibiotics
* No other concurrent experimental medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2001-07; Primary Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
MTD defined as the highest dose level at which =< 1/6 subjects experience a study related dose-limiting toxicity (DLT) as assessed by CTC version 2.0 | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Mary Cianfrocca, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States